CLINICAL TRIAL: NCT03339375
Title: The Effect of Esophageal Doppler Guided Goal-directed Hemodynamic Therapy
Brief Title: The Effect of Esophageal Doppler Guided Goal-directed Hemodynamic Therapy in Severe Trauma Patients
Acronym: GDT
Status: Completed | Type: Observational
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, In-kyong Yi, Clinical assistant professor, Ajou University School of Medicine
Other Study IDs: MED-OBS-17-314
Record Dates: First submitted 2017-11-05; First posted 2017-11-13 (Actual); Last update posted 2019-10-28 (Actual); Status verified 2019-10

CONDITIONS: Trauma
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- control: Monitoring arterial pressure, central venous pressure and pulse pressure variation
- esophagela Doppler: Monitoring arterial pressure, central venous pressure Insertion of esophageal Doppler probe to patient Monitoring stroke volume, cardiac output, corrected flow time from esophageal Doppler Use stroke volume optimization goal directed therapy protocol
  Interventions: Device: esophageal Doppler

INTERVENTIONS:
Device: esophageal Doppler — Goal directed fluid therapy using dynamic parameters from esophageal Doppler
  Groups: esophagela Doppler

SUMMARY:
Prospective randomized clinical trial Compare the goal-directed fluid therapy using esophageal Doppler and classic fluid therapy

DETAILED DESCRIPTION:
Goal directed fluid therapy becomes issue for enhanced recovery after surgery. In goal directed therapy, dynamic parameters, like stroke volume and cardiac output, is important. Esophageal Doppler is one of device which provides dymanic parameters.

In severe trauma cases, the effect of goal directed therapy is not known yet. So the aim of this study is comparing the results of goal directed therapy using esophageal Doppler and conventional fluid therapy.

ELIGIBILITY:
Inclusion Criteria:

* Severe trauma patients who undergo general anesthesia
* Initial serum lactate level > 2mmol/L

Exclusion Criteria:

* Severe traumatic brain injury
* THoracic surgery
* Age < 19 years old
* Impending arrest or post CPR state
* Severe facial trauma

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Severe trauma patients
  : Injury severity score > 15
Sampling Method: Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Lactate | Immediate postoperative (=initial ICU admission)
  Unit is mmol/L Inclusion criteria is initial lactate > 2mmol/L. Whole hospital use same device and unit to measure lactate. In this study, POCT lactate won't be used.
  After surgical resuscitation, lactate level is independent predictor of survival, because it represents tissue oxygenation.

SECONDARY OUTCOMES:
Acute Physiology and Chronic Health Evaluation II (APACHE II) score | Immediate postoperative
  ICU patient scoring system, score from 0 to 71, higher scores correspond to more severe disease and a higher risk of death
Creatinine | Immediate postop
  Kidney function

CONTACTS AND LOCATIONS:
Overall Officials: In Kyong Yi, MD, Principal Investigator — Ajou University School of Medicine
Locations (1):
- Ajou university school of medicine, Suwon, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No